CLINICAL TRIAL: NCT00093093
Title: Randomized, Double-Blind, Multicenter Study to Compare the Safety and Efficacy of Viramidine to Ribavirin in Treatment-Naive Patients With Chronic Hepatitis C
Brief Title: Study of Viramidine to Ribavirin in Patients With Chronic Hepatitis C Who Are Treatment Naive
Acronym: VISER2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RNA003142-302
Record Dates: First submitted 2004-09-30; First posted 2004-10-04 (Estimated); Last update posted 2012-06-22 (Estimated); Status verified 2012-06

CONDITIONS: Chronic Hepatitis C
Keywords: Viramidine; Ribavirin; Valeant; Hepatitis C; Pegylated interferon alfa-2a
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — taribavirin; Ribavirin; peginterferon alfa-2a

INTERVENTIONS:
Drug: Viramidine
Drug: Ribavirin
Drug: pegylated interferon alfa-2a

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of viramidine to ribavirin in chronic hepatitis C patients who have never before received treatment.

DETAILED DESCRIPTION:
Compare the efficacy and safety of viramidine 600 mg twice a day (BID) versus ribavirin 1000/1200 mg/day, both drugs administered in combination with pegylated interferon alfa-2a to treatment-naive patients with chronic hepatitis C (CHC)

ELIGIBILITY:
Inclusion Criteria:

* Treatment-naive patients with compensated chronic hepatitis C.
* HCV RNA >2000 copies/mL (780 IU/mL) as determined by NGI SuperQuant serum HCV RNA quantification, with a lower limit of detection of 100 copies/mL (39 IU/mL).

Exclusion Criteria:

* Severe neuropsychiatric disorders
* History or clinical manifestations of significant metabolic, hematological, pulmonary, ischemic heart disease, significant or unstable heart disease, gastrointestinal, neurological, renal, urological, endocrine, ophthalmologic disorders including severe retinopathy, or immune mediated disease
* Pregnant or breast-feeding patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900
Dates: Start 2004-06; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
- Efficacy: Undetectable plasma HCV RNA (less than 100 copies/mL) at the end of the 24-week post-treatment follow-up period.
- Safety: The proportion of patients with hemoglobin less than 10 g/dL at any time during treatment or at least 2.5 g/dL drop from baseline.

SECONDARY OUTCOMES:
- Efficacy: Undetectable plasma HCV RNA at treatment week 24
- Efficacy: Undetectable or at least a 2-log drop from baseline at treatment weeks 12 and 24
- Safety: Monitoring of adverse events
- Safety: Monitoring of abnormal changes in laboratory parameters that are not disease-related

CONTACTS AND LOCATIONS:
Overall Officials: Ralph T. Doyle, Study Director — Bausch Health Americas, Inc.
Locations (100):
- United States (53):
  - University of Arizona, Tucson, Arizona
  - UCSF Fresno- Internal Medicine, Fresno, California
  - Keck School of Medicine, University of Southern California, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Orange Coast Medical Group, Newport Beach, California
  - University of California Davis Medical Center, Sacramento, California
  - Research and Education, Inc., San Diego, California
  - California Pacific Medical Center, San Francisco, California
  - University of California San Francisco, San Francisco, California
  - San Mateo Medical Center, San Mateo, California
  - University of Colorado Health Sciences Center, Denver, Colorado
  - Rocky Mountain Gastroenterology, Lakewood, Colorado
  - University of Connecticut, Farmington, Connecticut
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Bach and Godofsky, Bradenton, Florida
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Atlanta Academic Research Group, Atlanta, Georgia
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - University of Louisville, Louisville, Kentucky
  - Louisiana State University Memorial Hospital, New Orleans, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Johns Hopkins, Baltimore, Maryland
  - Johns Hopkins University Medical Center, Baltimore, Maryland
  - Maryland Digestive Disease Research, Laurel, Maryland
  - Future Care Studies/Northgate Medical, Springfield, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Bradley Freilich, MD, Kansas City, Missouri
  - Saint Louis University School of Medicine, St Louis, Missouri
  - Atlantic Gastroenterology Associates, Egg Harbor, New Jersey
  - Regional Clinical Research, Inc., Johnson City, New York
  - North Shore University Hospital, Manhasset, New York
  - Cabrini Medical Center, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Jacobi Medical Center, The Bronx, New York
  - Bronx VA Medical Center, The Bronx, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Digestive Health Specialists, Winston-Salem, North Carolina
  - Consultants for Clinical Research, Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Research Solutions (SMO), Tulsa, Oklahoma
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Radiant Research - Austin, Austin, Texas
  - University of Texas, Dallas, Texas
  - VA Medical Center, Houston, Texas
  - INOVA Fairfax Hospital, Annadale, Virginia
  - Kaiser Permanente Medical Center, Falls Church, Virginia
  - Hunter Holmes McGuire Medical Center, Richmond, Virginia
  - Northwest Medical Specialties, Tacoma, Washington
- Argentina (5):
  - Hospital Italiano, Buenos Aires, Buenos Aires
  - Fundación CIDEA, Buenos Aires, Buenos Aires
  - Hospital Británico, Buenos Aires, Buenos Aires
  - Hospital Austral, Pilar, Buenos Aires
  - Hospital Centenario, Rosario, Santa Fe Province
- Australia (5):
  - Westmead Hospital, Westmead, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Royal Melbourne Hospital, Parkville, Victoria
  - The Alfred Hospital, Prahran, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Canada (4):
  - University of Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - University of Manitoba, Winnipeg, Manitoba
  - Toronto Western Hospital, Toronto, Ontario
- France (5):
  - CHU Grenoble Hôpital Michallon, Service d'Hépatogastroentérologie, Grenoble
  - Hopital Saint Joseph Service d'Hépato-gastroentérologie, Marseille
  - Hôpital de l'Archet 2 Service d'Hépato-Gastroentérologie, Nice
  - Hôpital Saint Antoine, Service d'Hépato-Gastroentérologie, Paris
  - C.H.U de Nancy - Hôpital de Brabois Adultes Service d'Hépato-gastroentérologie, Vandouevre Les Nancy
- Israel (3):
  - Rambam Medical Center Liver Unit, Haifa
  - Head of Liver Unit, Holy family Hospital, Nazareth
  - Tel Aviv Souraski Medical Center, Liver Unit, Department of Gastro-enterology, Tel Aviv
- Italy (5):
  - Malattie Infettive, Azienda Ospedaliera di Busto Arsizio, Busto Arsizio
  - Az. Osp. Universitaria Policlinico "Paolo Giaccone", Palermo
  - IRCCS Policlinico San Matteo, Pavia
  - Istituto Nazionale per le Malattie Infettive "Lazzaro Spallanzani" IRCCS, Rome
  - Divisione di Gastroenterologia, Azienda Ospedaliera S.Giovanni Battista, Torino
- Poland (6):
  - Wojewodzki Szpital Obserwacyjno-Zakazny im. T. Browicza, Bydgoszcz
  - Szpital Specjalistyczny, Chorzów
  - Katedra Chorob Zakaznych i Hepatologii Collegium Medicum Uniwersytetu Jagiellonskiego, Krakow
  - Katedra i Klinika Chorob Zakaznych Pomorskiej Akademii Medycznej, Szczecin
  - Klinika Chorob Wewnetrznych i Reumatologii CSK MON WIM, Warsaw
  - Wojewodzki Szpital Zakazny, Warsaw
- Fundacion de Investigacion de Diego, Santurce, Puerto Rico
- Russia (6):
  - Russian State Medical University, Moscow
  - City Hospital of Infectious Diseases #10, Saint Petersburg
  - Department of gastroenterology, Russian Military Academy; Regional Military Clinical Hospital №442, Saint Petersburg
  - City Hospital of Infectious Diseases #30, Saint Petersburg
  - Department of infectious diseases, Russian Military Academy, Saint Petersburg
  - Smolensk Medical Academy, Smolensk
- Spain (5):
  - Hospital Universitario Germans Trias i Pujol, Badalona
  - Hospital Santa Creu I Sant Pau, Barcelona
  - Hospital Universitario La Princesa, Madrid
  - Hospital Carlos III, Madrid
  - Hospital General Universitario de Valencia, Valencia
- United Kingdom (2):
  - Liver and Hepatobiliary Unit, Queen Elizabeth Hospital, Birmingham
  - Liver Unit, Royal Infirmary of Edinburgh, Edinburgh